CLINICAL TRIAL: NCT02377336
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Parallel Study of GS-6615 in Subjects With Chronic Stable Angina and Coronary Artery Disease
Brief Title: GS-6615 in Adults With Chronic Stable Angina and Coronary Artery Disease
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Anticipated recruitment challenges
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-279-1503; 2014-003994-41 (EudraCT Number)
Record Dates: First submitted 2015-02-26; First posted 2015-03-03 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Ischemic Heart Disease
Keywords: GS-6615; coronary heart disease; angina pectoris; late sodium current; myocardial ischemia; coronary artery disease; chronic stable angina
MeSH Terms: conditions — Myocardial Ischemia; Coronary Disease; Angina Pectoris; Coronary Artery Disease; Angina, Stable | interventions — eleclazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GS-6615 (Experimental): GS-6615 30 mg (5 x 6 mg) on Day 1, followed by 6 mg twice daily
  Interventions: Drug: GS-6615
- Placebo (Placebo Comparator): Placebo to match GS-6615 (5 tablets) on Day 1, followed by placebo to match GS-6615 twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GS-6615 — GS-6615 tablets administered orally
  Arms: GS-6615
Drug: Placebo — Placebo to match GS-6615 tablets administered orally
  Arms: Placebo

SUMMARY:
This study will evaluate the effect of GS-6615 in adults with chronic stable angina and coronary artery disease (CAD) receiving a stable daily dose of up to 2 antianginal medications. The study will consist of two periods: a 1 to 3 week Qualifying Period and a Treatment Period lasting 13 days (± 3 days). During the Qualifying Period and at the end of the Treatment Period, participants will undergo exercise tolerance testing.

ELIGIBILITY:
Inclusion Criteria:

* Able to perform a standardized treadmill exercise protocol
* At least a 3 month history of chronic stable angina triggered by physical effort and relieved by rest and/or short-acting nitroglycerin
* Coronary artery disease (CAD) documented by one or more of the following:

  * Angiographic evidence (either invasive or noninvasive) of ≥ 50% stenosis of one or more major coronary arteries
  * History of myocardial infarction (MI) documented by positive creatine kinase-myocardial band (CK-MB) enzymes, troponins, or electrocardiogram (ECG) changes
  * Noninvasive imaging stress test diagnostic of CAD (eg, nuclear perfusion scan, stress echocardiogram, stress cardiac magnetic resonance scan)
* Stable antianginal treatment with up to 2 antianginal agents

Exclusion Criteria:

* Inability to exercise or having exercise limitation due to other co-morbidities that may interfere with ability to perform required exercise tolerance testing (ETT)
* Presence of electrocardiographic or other abnormalities that interfere with ECG interpretation or may cause a false positive stress test
* History of heart failure as defined by New York Heart Association Class III-IV and/or known left ventricular ejection fraction ≤ 45%
* History of severe disabling angina as defined by Canadian Cardiovascular Society Class IV
* Myocardial infarction, acute coronary syndrome or coronary revascularization within 3 months prior to screening, or planned coronary revascularization during the study period
* Stroke or transient ischemic attack within 6 months prior to screening
* Chronic persistent atrial fibrillation
* Uncontrolled hypertension (seated systolic blood pressure (SBP) > 160 mm Hg or diastolic blood pressure (DBP) > 110 mm Hg)
* Body mass index (BMI) ≥ 36 kg/m^2

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-05; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in time to 1 mm ST-segment depression | Baseline; Day 13 (± 3 days)
  For treadmill-related endpoints, baseline is defined as the value derived from the last exercise tolerance testing performed during the qualifying period.

SECONDARY OUTCOMES:
Change from baseline in total exercise duration at the end of the double-blind treatment period | Baseline; Day 13 (± 3 days)
Time to onset of angina during exercise tolerance testing at the end of the double-blind treatment period | Baseline; Day 13 (± 3 days)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Yue, MD, Study Director — Gilead Sciences